CLINICAL TRIAL: NCT02220075
Title: Fiberoptic Evaluation of the LMA(Laryngel Mask Airway) Position During Anesthesia With Spontaneous Respiration or Controlled Ventilation in Children
Status: Completed | Type: Observational
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Other Study IDs: 4-2013-0550
Record Dates: First submitted 2014-08-14; First posted 2014-08-19 (Estimated); Last update posted 2019-03-26 (Actual); Status verified 2018-04

CONDITIONS: Pediatric Urologic Surgery
Keywords: fiberoptic, LMA, caudal block

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- spontaneous group: maintain spontaneous breathing during the operation, and recording tidal volume, ET CO2, respiratory rate, peak airway pressure, SpO2
- controlled group: controlled ventilation(tidal volume 8ml/kg, ET CO2 35~40mmHg) during the operation, recording peak airway pressure, SpO2

SUMMARY:
LMA(Laryngel Mask Airway) is useful for pediatrics surgery, and there are various methods of LMA insertion. When the investigators evaluate the LMA position, the investigators can use fiberoptic bronchoscope (Grade 1 to 4). For pediatric patients, clinical signs(airway pressure<20cmH2O, expiratory CO2 level)are seen normal but the grade is 3 or 4. And this will bring high risk of aspiration. Recent studies reported the LMA position after general anesthesia induction not after operation. Therefore, the investigators will observe the LMA position three times; after general anesthesia induction, after caudal block, and after operation as well as the difference regarding to spontaneous and controlled ventilation.

ELIGIBILITY:
Inclusion Criteria:

1. ASA physical status 1 or 2,
2. pediatric patients from 1month to 7 years old
3. under general anesthesia using LMA
4. getting informed consent from the guardian

Exclusion Criteria:

1. difficult airway
2. airway diseases ; URI, asthma, pneumonia
3. not getting informed consent from the guardian

Ages: 1 Month to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Pediatric patients who are planed to get urologic surgery under general anesthesia using LMA
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2015-03-04 (Actual); Primary Completion 2015-04-03 (Actual); Study Completion 2015-04-03 (Actual)

PRIMARY OUTCOMES:
sucess rate of LMA insertion | 1 hour

SECONDARY OUTCOMES:
FOB(fiberoptic bronchoscope) grading of LMA position | 1 hour
  Grade 1: only the larynx visible, Grade 2: larynz and epiglottis visible, Grade 3: epiglottis was impinging on the LMA grille, Grade 4: epiglottis was downfolded and the larynx could not be seen)

CONTACTS AND LOCATIONS:
Locations (1):
- Severance Hospital, Seoul, South Korea